CLINICAL TRIAL: NCT04679545
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Using Cannabidiol for the Treatment of Painful Diabetic Peripheral Neuropathy of the Feet
Brief Title: Using Cannabidiol to Treat Diabetic Peripheral Neuropathy of the Feet
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pure Green (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-DPN-20WS-2020
Record Dates: First submitted 2020-12-10; First posted 2020-12-22 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Cannabidiol; CBD; DPN; Diabetic Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: There are 2 groups in this trial: interventional group (active drug) and control group (placebo).
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized at a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD (Experimental): Subject will receive a 28-day supply of 20 mg CBD sublingual tablets to be taken 3 times a day for 28 days.
  Interventions: Drug: CBD
- Placebo Control (Placebo Comparator): A placebo sublingual tablet to be taken three times a day for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBD — A water-soluble sublingual tablet containing 20 mg of CBD.
  Arms: CBD
Drug: Placebo — An inactive compound.
  Arms: Placebo Control

SUMMARY:
The purpose of the study is to evaluate whether PG-DN-20WS is a better pain reliever in patients with diabetic neuropathic pain of the feet than a placebo.

DETAILED DESCRIPTION:
Subjects will be enrolled in the study for a maximum of 43 days, including an optional 14-day screening period, 28 days of active product administration, and followed by a post-treatment follow-up within 1 day.

The primary objective of this study is:

* To evaluate the safety of PG-DN-20WS for the treatment of painful DPN of the feet compared to a placebo control, including emergence of suicidal thoughts.

The secondary objectives of this study are:

* To evaluate the impact of PG-DN-20WS on subject's neuropathic pain, anxiety, and sleep quality compared to a placebo control.
* To evaluate the impact of PG-DN-20WS on the subject's impression of their response to the treatment compared to a placebo control.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 21 years of age;
2. Subject has a diagnosis of diabetic neuropathic pain of the feet determined by the subject's primary care physician or related health care provider.
3. Subject has a mean pain scale score of ≥ 5 recorded in the 7 days prior to randomization.
4. If female, the subject is postmenopausal (> 1 year), surgically sterile (> 3 months), had a hysterectomy, or is currently using 2 effective forms of birth control.
5. Subject has not taken marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and agrees to not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study.
6. If subject is currently taking gabapentin, pregabalin, or duloxetine, subject must be willing to and completes a 7-day washout of these medications prior to randomization.
7. Subject has not taken any NSAIDs and/or acetaminophen for at least 2 days prior to randomization.
8. Subject is willing to provide his/her written informed consent to participate in the study as stated in the informed consent document.
9. Subject is willing to use an electronic diary to enter trial information for 29 days.

Exclusion Criteria:

1. Subject is pregnant or lactating;
2. Subject has an allergy to cannabis, the Cannabaceae plant family (e.g., hemp, hops), palmitoylethanolamide, or terpenes;
3. Subject has a known allergy to active or inert ingredients of the investigational product;
4. Subject is taking a concomitant medication or treatment that would complicate use or interpretation of the study drug's effects (examples include: Cannabis or any cannabinoid products; Any drug or herbal product that influences the endocannabinoid system (ECS));
5. Subject is taking marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD for at least 14 days prior to this study, and does not promise that they will not take marijuana (cannabis) in any form, chemicals or extracts or foods or beverages or topical creams, lotions, gels, patches containing marijuana (cannabinoids, or and cannabis derivatives) including synthetic marijuana and/or CBD while participating in this study;
6. Subject currently resides in the state of Nebraska, Idaho, Iowa, or South Dakota.
7. Subject is currently being treated with antibiotics for sinus, throat, or lung infections;
8. Subject has shortness of breath associated with allergies;
9. Subject has uncontrolled asthma;
10. Subject has a fever and/or productive cough;
11. Subject has unstable angina, uncontrolled hypertension;
12. Subject currently or has a history of congestive heart failure;
13. Subject has any other unstable medical condition;
14. Subject has a personal or family history of schizophrenia;
15. Subject has a personal history or currently has suicidal ideation or attempted suicide;
16. Subject has a major neurological disorder, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, history of traumatic brain injury/head injury, and seizures.
17. Subject has taken pharmaceutical pain medicine of any kind, or has taken a NSAID and/or acetaminophen, within 2 days of randomization.
18. Subject has taken gabapentin, pregabalin, or duloxetine within 7 days prior to randomization or is unwilling to stop these medications.
19. Subject has an allergy to, or has an intolerance to, NSAIDs or acetaminophen.
20. Subject is currently taking any form of opioids.
21. Subject has a history of substance or alcohol abuse.
22. Subject has clinically significant illness, including cardiovascular disorders.
23. Subject has any condition in which the investigator believes will confound the data of the study or could put the subject at risk of harm.
24. Subject does not have access to a smart phone or does not know how to use a smart phone application.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | Four Weeks
  To evaluate the safety of PG-DN-20WS for the treatment of painful DPN of the feet compared to a placebo control assessed by Common Terminology Criteria For Adverse Events (CTCAE) v4.0.

SECONDARY OUTCOMES:
Pain as assessed by Numerical Pain Rating Scale (NPRS) | Four Weeks
  To evaluate the impact of PG-DN-20WS on the subject's neuropathic pain as assessed by utilizing a Numeric Pain Rating Scale (NPRS). NPRS is from 0-10, where higher scores indicate worse pain and lower scores indicate less pain reported by the subject.
Anxiety as assessed by the Zung Self-Rating Anxiety Scale (SAS) | Four Weeks
  To evaluate the impact of PG-DN-20WS on the subject's anxiety as assessed by the Zung Self-Rating Anxiety Scale (SAS). Subjects are given scores from 1-4 based on their responses to the survey, where a higher global score indicates a more severe form of anxiety and a lower global score indicates either a less severe form of anxiety or no anxiety presented by the subject.
Sleep Quality as assessed by Pittsburgh Sleep Quality Index (PSQI) | Four Weeks
  To evaluate the impact of PG-DN-20WS on the subject's anxiety as assessed by the Pittsburgh Sleep Quality Index (PSQI). Subjects are given scores from 0-3 based on their responses to the survey, where a higher global score indicates poor sleep quality and a lower global score indicates good sleep quality reported by the subject.
Subject's Response to Treatment as assessed by Patient's Global Impression of Change (PGIC) | Four Weeks
  To evaluate the impact of PG-DN-20WS on the subject's impression of their response to the treatment compared to a placebo control as assessed by Patient's Global Impression of Change (PGIC). Subjects indicate their overall impression of their response to treatment on 0-10 scale, where a higher number represents the subject feeling worse than before the intervention, and a lower number represents the subject feeling better than before the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kimless, M.D., Principal Investigator — Pure Green Pharmaceuticals
Locations (1):
- Pure Green Pharmaceuticals, Bloomfield Township, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quattrini C, Tesfaye S. Understanding the impact of painful diabetic neuropathy. Diabetes Metab Res Rev. 2003 Jan-Feb;19 Suppl 1:S2-8. doi: 10.1002/dmrr.360. PMID 12577252
- [Background] Callaghan BC, Cheng HT, Stables CL, Smith AL, Feldman EL. Diabetic neuropathy: clinical manifestations and current treatments. Lancet Neurol. 2012 Jun;11(6):521-34. doi: 10.1016/S1474-4422(12)70065-0. Epub 2012 May 16. PMID 22608666
- [Background] Argoff CE, Cole BE, Fishbain DA, Irving GA. Diabetic peripheral neuropathic pain: clinical and quality-of-life issues. Mayo Clin Proc. 2006 Apr;81(4 Suppl):S3-11. doi: 10.1016/s0025-6196(11)61474-2. PMID 16608048
- [Background] Sadosky A, Mardekian J, Parsons B, Hopps M, Bienen EJ, Markman J. Healthcare utilization and costs in diabetes relative to the clinical spectrum of painful diabetic peripheral neuropathy. J Diabetes Complications. 2015 Mar;29(2):212-7. doi: 10.1016/j.jdiacomp.2014.10.013. Epub 2014 Nov 8. PMID 25498300
- [Background] Gordois A, Scuffham P, Shearer A, Oglesby A, Tobian JA. The health care costs of diabetic peripheral neuropathy in the US. Diabetes Care. 2003 Jun;26(6):1790-5. doi: 10.2337/diacare.26.6.1790. PMID 12766111
- [Background] Singh R, Kishore L, Kaur N. Diabetic peripheral neuropathy: current perspective and future directions. Pharmacol Res. 2014 Feb;80:21-35. doi: 10.1016/j.phrs.2013.12.005. Epub 2013 Dec 25. PMID 24373831
- [Background] Boulton AJ: Management of Diabetic Peripheral Neuropathy. Clinical Diabetes. 2005;23(1):9-15.
- [Background] Wallace MS, Marcotte TD, Umlauf A, Gouaux B, Atkinson JH. Efficacy of Inhaled Cannabis on Painful Diabetic Neuropathy. J Pain. 2015 Jul;16(7):616-27. doi: 10.1016/j.jpain.2015.03.008. Epub 2015 Apr 3. PMID 25843054
- [Background] Bridges D, Ahmad K, Rice AS. The synthetic cannabinoid WIN55,212-2 attenuates hyperalgesia and allodynia in a rat model of neuropathic pain. Br J Pharmacol. 2001 Jun;133(4):586-94. doi: 10.1038/sj.bjp.0704110. PMID 11399676
- [Background] De Vry J, Denzer D, Reissmueller E, Eijckenboom M, Heil M, Meier H, Mauler F. 3-[2-cyano-3-(trifluoromethyl)phenoxy]phenyl-4,4,4-trifluoro-1-butanesulfonate (BAY 59-3074): a novel cannabinoid Cb1/Cb2 receptor partial agonist with antihyperalgesic and antiallodynic effects. J Pharmacol Exp Ther. 2004 Aug;310(2):620-32. doi: 10.1124/jpet.103.062836. Epub 2004 May 12. PMID 15140913
- [Background] Abrams DI, Jay CA, Shade SB, Vizoso H, Reda H, Press S, Kelly ME, Rowbotham MC, Petersen KL. Cannabis in painful HIV-associated sensory neuropathy: a randomized placebo-controlled trial. Neurology. 2007 Feb 13;68(7):515-21. doi: 10.1212/01.wnl.0000253187.66183.9c. PMID 17296917
- [Background] Ware MA, Wang T, Shapiro S, Robinson A, Ducruet T, Huynh T, Gamsa A, Bennett GJ, Collet JP. Smoked cannabis for chronic neuropathic pain: a randomized controlled trial. CMAJ. 2010 Oct 5;182(14):E694-701. doi: 10.1503/cmaj.091414. Epub 2010 Aug 30. PMID 20805210
- [Background] Wilsey B, Marcotte T, Deutsch R, Gouaux B, Sakai S, Donaghe H. Low-dose vaporized cannabis significantly improves neuropathic pain. J Pain. 2013 Feb;14(2):136-48. doi: 10.1016/j.jpain.2012.10.009. Epub 2012 Dec 11. PMID 23237736
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- [Background] Johnson JR, Burnell-Nugent M, Lossignol D, Ganae-Motan ED, Potts R, Fallon MT. Multicenter, double-blind, randomized, placebo-controlled, parallel-group study of the efficacy, safety, and tolerability of THC:CBD extract and THC extract in patients with intractable cancer-related pain. J Pain Symptom Manage. 2010 Feb;39(2):167-79. doi: 10.1016/j.jpainsymman.2009.06.008. Epub 2009 Nov 5. PMID 19896326
- [Background] De Gregorio D, McLaughlin RJ, Posa L, Ochoa-Sanchez R, Enns J, Lopez-Canul M, Aboud M, Maione S, Comai S, Gobbi G. Cannabidiol modulates serotonergic transmission and reverses both allodynia and anxiety-like behavior in a model of neuropathic pain. Pain. 2019 Jan;160(1):136-150. doi: 10.1097/j.pain.0000000000001386. PMID 30157131